CLINICAL TRIAL: NCT02711098
Title: InterLeukine Ancillary Study of the Therapeutic Hypothermia After Nonshockable Cardiac Arrest Trial.
Brief Title: IL Ancillary Study of the Therapeutic Hypothermia After Nonshockable Cardiac Arrest Trial.
Acronym: IL-HYPERION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IL Ancillary Study of HYPERION
Record Dates: First submitted 2016-03-06; First posted 2016-03-17 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; hypothermia; critical care
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted controlled temperature between 32.5 and 33.5°C (Active Comparator): Patients will be placed in targeted temperature control between 32.5 and 33.5 ° C for 24 hours and then slowly rewarmed for targeted temperature control between 36.5 and 37.5 ° C for 24 hours.
  Interventions: Biological: Inflammatory biomarkers dosage "Hypothermia Arm"
- Targeted controlled temperature between 36.5 and 37.5°C (Placebo Comparator): Patients will be placed in targeted temperature control between 36.5 and 37.5 ° C for 48 hours.
  Interventions: Biological: Inflammatory biomarkers dosage "Normothermia Arm"

INTERVENTIONS:
Biological: Inflammatory biomarkers dosage "Hypothermia Arm" — There is 6 dosage of inflammatory biomarker per patient included: H0, H12, H24, H36, H48 and H72 during targeted temperature management between 33°C and 37°C.
  Arms: Targeted controlled temperature between 32.5 and 33.5°C
Biological: Inflammatory biomarkers dosage "Normothermia Arm" — There is 6 dosage of inflammatory biomarker per patient included: H0, H12, H24, H36, H48 and H72 during targeted temperature management at 37°C.
  Arms: Targeted controlled temperature between 36.5 and 37.5°C

SUMMARY:
Cardiac arrest is at present a major cause of mortality as well as a cause of disability for the surviving victims.In Europe, every year counts as 300,000 cardiac arrests responsible for 250,000 deaths. Thus, less than 20 % of patients discharged home with impaired quality of life associated with symptoms of tiredness, stress, anxiety. The prognosis is related to the initial cardiac rhythm present during the initiation of resuscitation. Recent progress in the improvement of mortality and neurological outcome has been achieved over the last decade thanks to the systematic implementation of a period of targeted temperature control between 32 and 34 ° C in patients who benefited from the realization of at least one electrical external shock.

There are theoretical and clinical arguments to think that achieving the same way a period of targeted temperature control between 32 and 34 ° C in patients treated for cardiac arrest with a non- shockable rhythm on arrival can also benefit from this procedure. However other arguments are against this hypothesis including an increase in the risk of infection , worsening of the patient's hemodynamic status with no benefit to him. To answer this question, we conduce a randomized multicenter study testing the potential improvement of neurological outcome through this procedure targeted temperature control between 32.5 and 33.5 ° C in these patients.

IL Ancillary Study of HYPERION Trial will determine impact on inflammatory biomarkers of two temperature target for targeted temperature management (33°C or 37°C) after cardiac arrest in non-shockable rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest in nonshockable rhythm and
* Glasgow Coma Scale score ≤8. In patients receiving sedative therapy at ICU admission, the Glasgow Coma Scale score assessed by the emergency physician just before sedative therapy initiation is used.
* Patient must be randomized in a center which participate in the ancillary study.

Exclusion Criteria:

* No-flow time >10 min (time from collapse to initiation of external cardiac massage);
* Low-flow time >60 min (time from initiation of external cardiac massage to return of spontaneous circulation).
* Major hemodynamic instability (defined as a continuous epinephrine or norepinephrine infusion at a flow rate >1 μg/Kg/min)
* Time from cardiac arrest to study inclusion >300 min
* Moribund patient
* Child C cirrhosis of the liver
* Age <18 years
* Pregnant or breastfeeding woman
* Correctional facility inmate
* Previous inclusion in another randomized clinical trial on cardiac arrest with day-90 neurological outcome as the primary endpoint
* Patient without health insurance
* Decision by the patient or next of kin to refuse the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Interleukine 6 level between H0 and H72 | 72 hours
  Comparing the production of interleukin 6 (inflammatory cytokine) during targeted temperature management at 33 or 37 °C after cardiac arrest in non-shockable rhythm when help arrived and before the injection of adrenaline. The analysis of the primary endpoint will be performed using an analysis of covariance, taking into account the basal value of interleukine 6. Necessary data will be pre-processed.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Lascarrou, MD, Study Chair — CHD Vendee
Locations (14):
- France (14):
  - Centre hospitalier d'Annecy, Annecy
  - Medical Intensive Care Unit, Clermond Ferrand
  - CHU Dijon, Dijon
  - Medical Surgical Intensive Care Unit, La Roche-sur-Yon
  - Medical Surgical Intensive Care Unit, Lens
  - Medical Surgical Intensive Care Unit, Limoges
  - Medical Surgical Intensive Care Unit, Montauban
  - Medical Intensive Care Unit, Nantes
  - CHU Orleans, Orléans
  - Medical Intensive Care Unit, Poitiers
  - Medical Surgical Intensive Care Unit, Rodez
  - Medical Surgical Intensive Care Unit, Saint-Brieuc
  - Medical Surgical Intensive Care Unit, St-Malo
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://sjtrem.biomedcentral.com/articles/10.1186/s13049-015-0103-5